CLINICAL TRIAL: NCT01514162
Title: Post-Approval Study Protocol of the St. Jude Medical Trifecta Valve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1003
Record Dates: First submitted 2012-01-17; First posted 2012-01-20 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Heart Valve Diseases
Keywords: Trifecta Valve
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trifecta Valve Group (Experimental): Subjects implanted with a Trifecta valve.
  Interventions: Device: Trifecta valve

INTERVENTIONS:
Device: Trifecta valve — surgical replacement of aortic valve

SUMMARY:
To further evaluate the long term clinical safety and effectiveness of the Trifecta valve

DETAILED DESCRIPTION:
To further evaluate the long term clinical safety and effectiveness of the Trifecta valve in subjects who had a Trifecta valve implanted during the IDE study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects implanted with a Trifecta valve at one of the US sites of the IDE study.
* Subject met eligibility criteria of IDE study
* Subject agrees to complete study follow-up visits
* Subject provides written informed consent

Exclusion Criteria:

* Subject currently participating in another device or drug study
* Subject unable or unwilling to return for study follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2012-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Abbott Northwestern Hospital Cardiac Surgical Associates, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Mission Hospital, Asheville, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt Heart Institute, Nashville, Tennessee
  - Intermountain Heart & Lung Surgical Associates, Murray, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trifecta Valve Group
Started | 245
Completed | 160
Not Completed | 85

BASELINE CHARACTERISTICS:
Arm/Group | Trifecta Valve Group
Number analyzed (Participants) | 245
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 172
Region of Enrollment [Number; unit: participants]
  United States | 245

OUTCOME MEASURES:

1. Primary Outcome: Late Adverse Event Incidence
Description: Late patient years are calculated from 31 days post-implant to the date of the last follow-up visits (or contact) or adverse events.
  Late Patient year calculation:[(Number of late adverse events/sum of late patient years) x 100]
Time Frame: 5 years
Measure: Number; unit: event/100-patient years
Arm/Group | Trifecta Valve Group
Number analyzed (Participants) | 245
event/100-patient years
  Thromboembolism | 7
  Valve thrombosis | 0
  Nonstructural Dysfunction | 0
  Structural Deterioration | 4
  Mortality | 9
  Endocarditis | 0

2. Secondary Outcome: Characterize Patient NYHA Functional Classification Status
Description: The New York Heart Association (NYHA) functional classification system relates symptoms to everyday activities and the patient's quality of life.
  Class I. Patients with cardiac disease but without resulting limitation of physical activity.
  Class II. Patients with cardiac disease resulting in slight limitation of physical activity. They are comfortable at rest.
  Class III. Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest.
  Class IV. Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of heart failure or the anginal syndrome may be present even at rest.
  The Criteria Committee of the New York Heart Association. Nomenclature and Criteria for Diagnosis of Diseases of the Heart and Great Vessels. 9th ed. Boston, Mass: Little, Brown & Co; 1994:253-256.
Time Frame: 5 years
Population: Number of participants analyzed is those subjects with a visit and completed assessment
Measure: Number; unit: participants
Arm/Group | Trifecta Valve Group
Number analyzed (Participants) | 189
participants
  NYHA I | 171
  NYHA II | 16
  NYHA III | 2
  NYHA IV | 0

3. Secondary Outcome: Report the Hemodynamic Performance of the Valve
Description: Gradient is the pressure difference from one side of the valve to the other side of the valve. For this study pressure is measured in mmHg.
  Mean gradient for each patient is the average of the pressure differences from one side of the valve to the other side of the valve.
  Mean gradient for each valve size (19mm, 21mm, 23mm, 25mm, 27mm, 29mm)is the average of the mean gradient for each patient with that valve size.
Time Frame: 5 years
Population: Aortic valve mean gradient at 5 years for participants analyzed with a visit and completed assessment
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Trifecta Valve Group
Number analyzed (Participants) | 176
mmHg
  19mm | 15.4 (5.9)
  21mm | 10.4 (5.6)
  23mm | 9.2 (4.9)
  25mm | 7.9 (3.7)
  27mm | 8.4 (8.8)
  29mm | 6.1 (2.3)

ADVERSE EVENTS:
Arm/Group | Trifecta Valve Group
Serious Adverse Events (participants affected / at risk) | 39/245
Other Adverse Events (participants affected / at risk) | 0/245
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trifecta Valve Group (N=245)
Thromboembolism (Cardiac disorders) | 9 (9)
Valve thrombosis (Cardiac disorders) | 0 (0)
Major bleed (Vascular disorders) | 24 (24)
Nonstructural dysfunction (Cardiac disorders) | 0 (0)
Endocarditis (Cardiac disorders) | 0 (0)
Clinically significant hemolysis (Blood and lymphatic system disorders) | 0 (0)
Structural deterioration (Cardiac disorders) | 4 (4)
Reoperation (Surgical and medical procedures) | 2 (2)
Valve related mortality (Cardiac disorders) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other